CLINICAL TRIAL: NCT02149745
Title: Effect of Calling the Patient's Name on Recovery From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JHSeo_Calling
Record Dates: First submitted 2014-05-08; First posted 2014-05-29 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Delayed Emergence From Anesthesia
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Calling the patient's name (Experimental): The anesthesiologist tries to recover the patient's consciousness by calling the patient's name
  Interventions: Procedure: Calling the patient's name
- Not calling the patient's name (Experimental): The anesthesiologist tries to recover the patient's consciousness by giving verbal stimulus other than the patient's name
  Interventions: Procedure: Not calling the patient's name

INTERVENTIONS:
Procedure: Calling the patient's name — calling the patient's name during anesthesia reversal
  Arms: Calling the patient's name
Procedure: Not calling the patient's name — giving verbal stimulus other than the patient's name during anesthesia reversal
  Arms: Not calling the patient's name

SUMMARY:
The purpose of this study is to find if we can shorten the recovery time by calling the patient's name during anesthesia reversal.

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 20-70
* patient receiving breast cancer surgery under general anesthesia with total intravenous anesthesia using remifentanil and propofol, and intubated with LMA

Exclusion Criteria:

* refusal of consent
* patients taking CNS stimulants
* general anesthesia with other agents than propofol and remifentanil
* intubated with other equipments than LMA
* chronic alcoholic patient
* patients with convulsive disorder

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Difference in recovery time between the two groups | 1 min,2 min,3 min, 4min, 5min, 6min, 7min, 8min, 9min, 10min after stopping injection of anesthetics
  difference in recovery time (eye opening time, extubation time) after stopping injection of anesthetics, and the time when the patient's bispectral index value displayed on the monitor is above 60

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea